CLINICAL TRIAL: NCT05829018
Title: Elucidating the High Cardiovascular Disease Risk in South Asians: Focus on Monocyte Phenotype and Incretin Hormones
Brief Title: Elucidating the High Cardiovascular Disease Risk in South Asians
Acronym: CAMI
Status: Unknown | Phase: Not Applicable | Type: Interventional
Last Known Status: Recruiting
Sponsor: Leiden University Medical Center (Other)
Responsible Party: Principal Investigator, mrboon, Mariëtte Boon, MD PhD, Principal Investigator, Leiden University Medical Center
Allocation: Non-Randomized | Model: Parallel | Masking: Single | Purpose: Basic Science
Other Study IDs: 22097
Record Dates: First submitted 2023-03-18; First posted 2023-04-25 (Actual); Last update posted 2023-04-25 (Actual); Status verified 2023-04

CONDITIONS: Cardiovascular Diseases
MeSH Terms: conditions — Cardiovascular Diseases

STUDY DESIGN:
Intervention Model Description: Cross-sectional study
Who Masked: Participant
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (4):
- Dutch South Asian males (Active Comparator): males of Dutch South Asian descent, as defined as having 4 grandparents that originally descended from either Surinam, Bangladesh, India, Nepal, Pakistan, Afghanistan, Bhutan or Sri Lanka
  Interventions: Diagnostic Test: Mixed meal test
- Dutch South Asian females (Active Comparator): females of Dutch South Asian descent, as defined as having 4 grandparents that originally descended from either Surinam, Bangladesh, India, Nepal, Pakistan, Afghanistan, Bhutan or Sri Lanka
  Interventions: Diagnostic Test: Mixed meal test
- Dutch Europid males (Active Comparator): males of Europid descent, as defined as having 4 grandparents from European origin
  Interventions: Diagnostic Test: Mixed meal test
- Dutch Europid females (Active Comparator): females of Europid descent, as defined as having 4 grandparents from European origin
  Interventions: Diagnostic Test: Mixed meal test

INTERVENTIONS:
Diagnostic Test: Mixed meal test — Nutridrink 270 mL 405 kcal, 49 Energy% carbohydrates, 35 Energy% fat, 16 Energy% protein, vitamins, and minerals
  Other Names: Nutridrink, Nutricia

SUMMARY:
The goals of this cross-sectional study are to compare immune cell composition and release of incretin hormones following a meal in healthy Dutch South Asians and Dutch Europids. The primary aim is to assess potential differences between Dutch South Asians and Dutch Europids with respect to immune cell composition and monocyte phenotype.

The secondary aim is to assess potential differences between Dutch South Asians and Dutch Europids with respect to hunger and satiety hormones following a mixed meal test.

The investigators will include healthy lean male and female participants of Dutch South Asian and Dutch Europid descent (n=48 in total).

DETAILED DESCRIPTION:
Rationale:

The worldwide increasing incidence of type 2 diabetes mellitus (T2DM) and cardiovascular diseases (CVD) has significant health and economic implications. Interestingly, the vulnerability to develop CVD is higher in Dutch South Asians (from here on called: South Asians) than in Dutch Europids. Several factors are suspected to contribute to this high CVD risk in South Asians, including higher prevalence of central obesity, insulin resistance and dyslipidemia as well as lifestyle factors such as lower amount of exercise and consumption of a diet high in ultra-processed foods. The higher susceptibility to develop central obesity and insulin resistance in the South Asian population would fit with increased sensitivity of the glucocorticoid receptor (GR) compared with Europids, resulting in increased activity of the glucocorticoid system. Furthermore, dyslipidemia and inflammation are central risk factors for the development of atherosclerosis, the most important driver of CVD. Levels of C-reactive protein (CRP), a non-specific marker for low-grade inflammation in the body, were shown to be higher in South Asians compared to Dutch Europids already just after birth. The fact that CRP levels are already higher in South Asian neonates suggests that genetic susceptibility may underlie the pro-inflammatory phenotype of South Asians. Up till now, only little is known about the regulation of the immune system of South Asians. Moreover, the phenotype of monocytes, the immune subset that plays a central role in atherosclerosis development, has also not been studied in South Asians so far. In addition, the underlying cause for the more proinflammatory phenotype is currently unknown in South Asians. Since this susceptibility further aggravates their high CVD risk, it is important to be further uncovered. Incretin hormones (glucagon-like peptide-1 (GLP-1) and glucose-dependent insulinotropic polypeptide (GIP)), secreted by intestinal cells following a meal, have direct anti-inflammatory effects and the incretin system has not been studied in detail in South Asians compared to Europids. Considering their high CVD risk, it is hypothesized that Dutch South Asians have a relatively pro-inflammatory balanced immune system including more pro-inflammatory monocytes compared with Dutch Europids and a lower release of anti-inflammatory incretin hormones following a meal, further contributing to their proinflammatory phenotype. Moreover, we hypothesize increased GR sensitivity in Dutch South Asians compared with Dutch Europids, contributing to their disadvantageous metabolic phenotype.

Objectives:

Primary objectives

1. To compare immune cell composition between lean adolescent Dutch South Asian and BMI- and age-matched Dutch Europids
2. To compare the monocyte phenotype between lean adolescent Dutch South Asian and BMI and age-matched Dutch Europids
3. To compare functional and metabolic characteristics of monocytes between lean adolescent Dutch South Asian and BMI- and age-matched Dutch Europids Secondary objectives
4. To compare GR sensitivity between lean adolescent Dutch South Asian and BMI- and age-matched Dutch Europids
5. To compare the release of incretins (GLP-1 and GIP) during a mixed meal tolerance test (MMTT) between lean adolescent Dutch South Asian and BMI- and age-matched Dutch Europids
6. To compare markers of glucose metabolism (glucose, insulin) during an MMTT between lean adolescent Dutch South Asian and BMI- and age-matched Dutch Europids
7. To compare markers of lipid metabolism (e.g. free fatty acids (FFA), triglycerides (TG), high-density-lipoprotein (HDL), total cholesterol) during an MMTT between lean adolescent Dutch South Asian and BMI- and age-matched Dutch Europids

Study design:

This study is a cross-sectional study carried out at the Leiden University Medical Centre (LUMC). The study encompasses one screening phone call and half a study day that takes approximately 4.5 hours per participant.

Study population:

The study will be carried out in Dutch South Asian men (n=12) and Dutch South Asian women (n=12) with a body mass index (BMI) between 18 and 23 kg/m2 and aged 18-30 years and BMI- and age-matched Dutch European men (n=12) and women (n=12); 48 participants in total.

Main study parameters/endpoints:

Differences between Dutch South Asians and Dutch Europids with respect to:

* Immune cell composition (flow cytometry)
* Monocyte phenotype, including activation markers and receptors (flow cytometry)
* Functional and metabolic characteristics of monocytes (in vitro stimulation with lipopolysaccharide (LPS), GLP-1 and GIP and Seahorse measurements to assess substrate use of monocytes)
* Release of incretin hormones (GLP-1 and GIP) following an MMTT
* GR sensitivity (bioassay in mononuclear cells and hair cortisol)

Clinical implications:

The results of this study may improve understanding of the predisposition of South Asians to CVD. More specifically, on the one hand the focus will be on the inflammatory processes that are involved including the monocyte phenotype of South Asians. Besides, the investigators will study whether a disturbed release of the incretin hormones GLP-1 and GIP may contribute to the proinflammatory phenotype of South Asians and whether in South Asians increased GR sensitivity is present. Eventually, the results of this study might reveal opportunities for medical intervention in South Asians focused on reducing inflammation (e.g. incretin-based therapy), resulting in early prevention of CVD.

Nature and extent of the burden and risks associated with participation, benefit, and group relatedness:

Participants will neither directly nor personally benefit from participating in this research project. At the same time, no large side effects are expected when taking part in this study. After informed consent, anthropometric measures will be taken, venous blood (130.5 mL) will be drawn for investigating the above-mentioned objectives and an MMTT will be performed to assess release of incretin hormones and insulin sensitivity. All measurements will be done in one study day that takes approximately 4.5 hours per participant.

ELIGIBILITY:
Inclusion Criteria:

* Biologically male and female
* South Asian or Dutch European ethnicity (South Asian ethnicity is defined as having 4 grandparents that originally descended from either Surinam, Bangladesh, India, Nepal, Pakistan, Afghanistan, Bhutan or Sri Lanka)
* Age from 18 to 30 years old
* BMI 18-23 kg/m2
* Capable of giving written informed consent
* Able to comply with the requirements and restrictions listed in the informed consent form

Exclusion Criteria:

* (auto-) immune disease(s) including type 1 or 2 diabetes mellitus, chronic kidney disease, hepatic disease, inflammatory bowel disease, thyroid disease and rheumatoid arthritis.
* Genetic lipid-associated disorders such as familial hypercholesterolemia
* Any chronic renal or hepatic disease
* Use of medication known to influence glucose and/or lipid metabolism (e.g. beta-blockers, antidepressants, corticosteroids)
* Abuse of alcohol or other substances
* Smoking
* Vigorous exercise (>3 times/week)
* Milk or soy allergy

Ages: 18 Years to 30 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult
Gender Based: Yes — Biologically male and female
Enrollment: 48 (Estimated)
Dates: Start 2023-04 (Estimated); Primary Completion 2024-03 (Estimated); Study Completion 2024-06 (Estimated)

PRIMARY OUTCOMES:
Immune cell composition | Baseline
  Differences in immune cell composition via flow cytometry in Dutch South Asians and Dutch Europids, via the measurement of CD14, CD16, HLA-DR (monocytes), CD3, CD4, CD8, CD46 and CD19
Monocyte phenotype | Baseline
  Differences in the monocyte phenotype via the measurements of monocyte subset percentage and their expression of key proteins, including inflammatory and anti-inflammatory markers and receptors via flow cytometry of fresh blood samples in Dutch South Asians and Dutch Europids.
  After red blood cell lysis, immune cells will be stained by a range of monocyte/immune/activation markers (e.g. CD14, CD16, CD80, CD86, HLA-DR, CCR2, CD11c, CD36, CX3CR1, CD45RA, CD206, CD200R), fixed and stored at 4°C for follow-up fluorescence-activated cell sorting (FACS).
Functional and Metabolic characteristics of monocytes | Baseline
  Difference in functional and metabolic characteristics of monocytes via in vitro stimulation with lipopolysaccharides, GLP-1 and GIP and Seahorse measurements in Dutch South Asians and Dutch Europids
  Whole blood will be activated in cell culture dishes in vitro with the prototypical pro-inflammatory Toll-like Receptor 4 trigger LPS with/without preincubation with GLP-1 and/or GIP and supernatant will be collected and stored at -80°C. Once samples from all donors are collected, the production of cytokines will be assessed (i.e. IL-6, TNF-α, IL-12p70, IL-8) by Enzyme-Linked Immune Sorbent Assay

SECONDARY OUTCOMES:
Incretin hormones | Baseline, and after 10, 20, 30, 60, 90, 120, 180 and 240 minutes after the mixed meal
  Difference in the release of hunger and satiety hormones in Dutch South Asians and Dutch Europids measured by the concentration of glucose, insulin, glucagon, GIP, GLP-1, leptin, ghrelin, CKK and PYY.
Glucocorticoid receptor sensitivity | Baseline
  In short, in PBMCs the trans-activation and trans-repression of four GR target genes (e.g. GILZ, FK506 binding protein 5, interleukin-2 and interleukin-6) in response to dexamethasone will be assessed using RT-qPCR, in addition to expression of several GR isoforms including the GRα, GRβ and GR-P. Furthermore, PBMCs will be stimulated with increasing concentrations of dexamethasone to determine the half maximum (EC50) and maximum effective concentration in addition to the half maximum (IC50) and maximum inhibitory concentration as a measure of GR sensitivity.

CONTACTS AND LOCATIONS:
Overall Officials: Mariëtte R Boon, Principal Investigator — Leiden University Medical Center
Locations (1):
- Leiden University Medical Center, Leiden, Netherlands

IPD SHARING:
Plan to Share IPD: No